CLINICAL TRIAL: NCT03591029
Title: Evaluation of PCO2 and PO2 Values in the Pulmonary Artery and in the Superior Vena Cava: Relationship With Cardiac Output, Hematocrit and Post Operative Organ Dysfunction
Brief Title: Evaluation of PCO2 and PO2 Values in the Pulmonary Artery and Superior Vena Cava
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Franco Cavaliere, Professor, Catholic University of the Sacred Heart
Other Study IDs: Polm01
Record Dates: First submitted 2018-07-02; First posted 2018-07-18 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood samples — blood samples will be obtained from the superior vena cava (via centra venous catheter), from the pulmonary artery (via Swan Ganz catheter), and from a radial or femoral artery catheter

SUMMARY:
The study is about comparing blood samples obtained from the superior vena cava and the pulmonary artery. The investigators will compare the values of PCO2 and PO2 from these two sites, in order to see if exists a PCO2 gap and a PO2 gap, different from zero. Moreover the investigators want to find out if these gaps are related with changes in the cardiac output, the hematocrit or if they can predict post operative dysfunctions.

Blood samples will be taken at six different times as scheduled by the protocol. Along with the two venous blood samples, an arterial blood sample will be taken too, from a radial of femoral artery catheter.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* patient undergoing cardiac surgery with extracorporeal circulation
* hemodynamic monitoring with a central venous catheter and a Swan Ganz catheter placed in the internal left giugulare vein

Exclusion Criteria:

* severe tricuspid insufficiency
* EF < 50%
* SOFA score >1 in at least one of all the criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Will be enrolled adult patients only , eligible for cardiac surgery (CABG, valvular replacement, aortic surgery) with extra corporeal circulation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
PCO2 gap changes | two days
  See if exists a PCO2 pa-svc gap different from zero in patients undergoing cardiac surgery
PO2 gap changes | two days
  See if exists a PCO2 pa-svc gap different from zero in patients undergoing cardiac surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - catholic University of the sacred Heart, Rome
  - Francesca Bevilacqua, Rome

IPD SHARING:
Plan to Share IPD: No